CLINICAL TRIAL: NCT02550496
Title: Evaluation of Trichoscopy in the Diagnosis of Tinea Capitis. Prospective, Multicenter Study (ETDT)
Brief Title: Evaluation of Trichoscopy in the Diagnosis of Tinea Capitis
Acronym: ETDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2014_843_0019
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Dermoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tinea capitis (Experimental)
  Interventions: Device: Dermoscopy

INTERVENTIONS:
Device: Dermoscopy
  Other Names: Trichoscopy

SUMMARY:
Waiting for a proof by mycological culture is usually necessary before starting a systemic antifungal therapy. It therefore seems to us interesting to evaluate the benefit of using dermoscopy in clinical diagnosis of Tinea Capitis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinically diagnosed tinea capitis
* Patient has signed informed consent

Exclusion Criteria:

* Patient with kerion or tinea favosa
* Antifungal treatment within 15 days prior to inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
The presence of several hair with at least one dermoscopic appearance specific of tinea capitis | baseline
  The presence of several hair with at least one dermoscopic appearance Specific of tinea capitis ( corkscrew hair , comma hairs, interrupted (Morse code-like) hairs, hair shafts covered by whitish sheaths, zig-zag shaped hairs) correlating with The growth of a dermatophyte in the fungal culture.

SECONDARY OUTCOMES:
Dermoscopic appearance (corkscrew hair, comma hairs, interrupted (Morse code-like) hairs, hair shafts covered by whitish sheaths, zig-zag shaped hairs) according to microscopic pathogenic species. | baseline
Concordance of dermoscopic appearance for each of the two operators. | baseline
  Concordance between dermoscopic interpretation (corkscrew hair, comma hairs, interrupted (Morse code-like) hairs, hair shafts covered by whitish sheaths, zig-zag shaped hairs) of the dermatologist during the initial consultation and dermoscopic interpretation on the photographs by a blinded trained practitioner.
Presence of a green fluorescence or not under the light of a Wood's lamp by comparing it with the result of the fungal culture. | baseline
Introduction or not of a local or general presumptive treatment by the clinician while waiting for the result of the fungal culture. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lok, PU-PH, Principal Investigator — CHU Amiens, Service de Dermatologie
Locations (4):
- France (4):
  - CHU Amiens, Amiens, Picardie
  - CHU Caen, Caen
  - CHRU Lille, Lille
  - CHU Rouen, Rouen

REFERENCES:
- [Result] Zalaudek I, Argenziano G, Di Stefani A, Ferrara G, Marghoob AA, Hofmann-Wellenhof R, Soyer HP, Braun R, Kerl H. Dermoscopy in general dermatology. Dermatology. 2006;212(1):7-18. doi: 10.1159/000089015. PMID 16319467
- [Result] Micali G, Lacarrubba F, Massimino D, Schwartz RA. Dermatoscopy: alternative uses in daily clinical practice. J Am Acad Dermatol. 2011 Jun;64(6):1135-46. doi: 10.1016/j.jaad.2010.03.010. Epub 2011 Feb 3. PMID 21292346
- [Result] Ekiz O, Sen BB, Rifaioglu EN, Balta I. Trichoscopy in paediatric patients with tinea capitis: a useful method to differentiate from alopecia areata. J Eur Acad Dermatol Venereol. 2014 Sep;28(9):1255-8. doi: 10.1111/jdv.12246. Epub 2013 Aug 24. PMID 23980908
- [Result] Hughes R, Chiaverini C, Bahadoran P, Lacour JP. Corkscrew hair: a new dermoscopic sign for diagnosis of tinea capitis in black children. Arch Dermatol. 2011 Mar;147(3):355-6. doi: 10.1001/archdermatol.2011.31. No abstract available. PMID 21422348
- [Result] Sandoval AB, Ortiz JA, Rodriguez JM, Vargas AG, Quintero DG. [Dermoscopic pattern in tinea capitis]. Rev Iberoam Micol. 2010 Sep 30;27(3):151-2. doi: 10.1016/j.riam.2010.02.003. Epub 2010 Mar 24. No abstract available. Spanish. PMID 20346297
- [Result] Slowinska M, Rudnicka L, Schwartz RA, Kowalska-Oledzka E, Rakowska A, Sicinska J, Lukomska M, Olszewska M, Szymanska E. Comma hairs: a dermatoscopic marker for tinea capitis: a rapid diagnostic method. J Am Acad Dermatol. 2008 Nov;59(5 Suppl):S77-9. doi: 10.1016/j.jaad.2008.07.009. PMID 19119131